CLINICAL TRIAL: NCT01043796
Title: Malaria Transmission Consortium: The Added Effects of Insecticide Treated Materials, Artemisinin-containing Combination Treatments, and Larviciding on Malaria Transmission and Illness
Brief Title: Evaluation of Insecticide Treated Nets and Wall Liners for the Prevention of Malaria
Acronym: MTC-ITWL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCZVED-5794
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Malaria
Keywords: Insecticide treated wall liners; Insecticide treated nets; Incidence cohort
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insecticide treated nets and wall liners (Experimental)
  Interventions: Other: Insecticide treated nets and wall liners
- Insecticide treated nets alone (Active Comparator)
  Interventions: Other: Insecticide treated nets alone

INTERVENTIONS:
Other: Insecticide treated nets and wall liners — Participants will be provided a long-lasting insecticide treated net recommended by the WHO Pesticide Evaluation Scheme. Households where participants reside will be fitted with insecticide treated wall liners.
  Arms: Insecticide treated nets and wall liners
Other: Insecticide treated nets alone — Participants will be provided with a long-lasting insecticide treated net recommended by the WHO Pesticide Evaluation Scheme
  Arms: Insecticide treated nets alone

SUMMARY:
The purpose of this study is to determine whether insecticide treated wall liners, in combination with insecticide treated nets, reduce the incidence of malaria infections compared to insecticide treated nets alone.

DETAILED DESCRIPTION:
Insecticide treated nets (ITNs) have been shown to reduce malaria related morbidity and mortality and are increasingly being scaled up throughout sub-Saharan Africa. However, ITNs alone are unlikely to reduce transmission to zero in most settings and additional vector control tools are necessary. One new promising strategy is the use of insecticide treated wall liners (ITWLs). These are textiles treated with an insecticide that are used to line the inner walls of houses. The wall liners are considered a long-lasting alternative to indoor residual spraying which is also used for malaria vector control but is expensive to implement.

Within 6 pairs of villages, we plan to randomly allocate one village in each pair to receive either ITNs or ITNs plus ITWLs. Households will be randomly selected from each village and all children between the ages of 6 months and 11 years will be enrolled in a cohort study. The children will be cleared of existing infections and then followed monthly until they are found to be infected with malaria. The study will last for 6 months and will demonstrate whether the ITWLs provide additional protection against malaria over that provided by the use of ITNs.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months up to 11 years
* Living in the study area and remaining in the study area for the duration of the study
* Informed consent provided by parents

Exclusion Criteria:

* No informed consent
* Living outside the study area, or likely to move outside study area
* Severely ill and unlikely to be able to complete study

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1730 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Incidence of new malaria infections | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: John E Gimnig, Ph.D., Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Kenya Medical Research Institute, Kisumu, Nyanza, Kenya